CLINICAL TRIAL: NCT00968864
Title: A Phase II Study Using the CliniMACS® Device for CD34+ Cell Selection and T Cell Depletion for Graft-versus-Host Disease Prophylaxis in Alternative Donor Stem Cell Transplant Recipients
Brief Title: T-cell Depleted Alternative Donor Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor/ PI leaving institution, no plans to continue this research at this time
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCH BMT 09-01
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2017-10

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Chronic Myeloid Leukemia; Myelodysplastic Syndrome; Lymphomas; Bone Marrow Failure; Hemoglobinopathy; Immune Deficiency; Osteopetrosis
Keywords: T cell depleted; Matched unrelated donors; Haplocompatible donors
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Lymphoma; Bone Marrow Failure Disorders; Hemoglobinopathies; Immunologic Deficiency Syndromes; Osteopetrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CliniMACS® (T cell depletion) (Experimental): Recipients will receive T cell-depleted PBSC from eligible donors after receiving conditioning therapy using CliniMACS® device.
  Interventions: Device: CliniMACS® (T cell depletion)

INTERVENTIONS:
Device: CliniMACS® (T cell depletion) — Stem cells will be collected from donors after they receive Granulocyte colony-stimulating factor (G-CSF). The cells will be processed using the CliniMACS device to select for CD34+ stem cells and to deplete T cells. Recipients will receive conditioning therapy that is based on their disease type and then receive the CD34+ stem cells.
  Other Names: CliniMACS device; T-cell depletion

SUMMARY:
The primary purpose is to determine the ability of CD34+ selection and T cell depletion using the CliniMACS® device to prevent severe acute graft-versus-host disease (GVHD) in patients receiving a stem cell transplant from an alternative (unrelated and mismatched related) donor. The secondary objectives include evaluation of engraftment, immune recovery, and post-transplant infections.

Patients requiring stem cell transplants for either malignant (cancerous) or non-malignant disease will be included in the study. The recipients will be grouped into one of two groups based on whether the donor is mismatched related (Cohort A) or unrelated (Cohort B). The patient will receive a conditioning regimen including chemotherapy drugs and/or total body irradiation based on the disease for which the transplant is performed.

DETAILED DESCRIPTION:
A major issue in alternative donor (mismatched related and unrelated donor transplantation is the development of graft-versus-host disease (GVHD). Several clinical trials have shown that the use of T-cell depleted peripheral blood stem cells (PBSC) reduces GVHD in alternative donor transplants. The purpose of this study is to determine the ability of CD34 positive selection and T cell depletion using the CliniMACS® Device as the only GVHD prophylaxis to prevent severe acute GVHD in recipients of an alternative donor PBSC transplant. Mismatched related donors will match at least 3 of 6 Human leukocyte antigens(HLA)(haplocompatible) and unrelated donors will match at least 6 out of 8 HLA antigens with the transplant recipient. The conditioning therapy including chemotherapy, anti-thymocyte globulin (ATG), +/- total body irradiation (TBI) will be based on the patient's diagnosis. The transplant recipient will be followed for 5 years after transplant for GVHD, engraftment, post-transplant infections, disease relapse, and overall survival. In addition, this study will serve as a platform for a companion study of therapy to accelerate immune recovery after transplant.

ELIGIBILITY:
Inclusion Criteria:

* Age < 30 years
* Patient must have a malignant or non-malignant disease that can benefit from alternative stem cell transplantation. Examples include acute and chronic leukemias, myelodysplastic syndrome, lymphoma, severe acquired and congenital cytopenias, white and red blood cell abnormalities, and immunodeficiencies.
* Patients with acute lymphoblastic leukemia must be in morphological remission (< 5% blasts) at the time of transplant. Patients with acute non-lymphocytic leukemia will preferably be in morphologic remission but may be enrolled when aplastic after chemotherapy or with < 20% blasts. Patients with lymphoma must be in complete or close to complete remission (if residual adenopathy, PET scan must be negative or only have slight uptake, eg. SUV < 2).
* Patients must lack a healthy HLA-identical related donor of at least one year of age.
* Patient must have a mismatched related or an unrelated donor who is:

  1. Able to receive G-CSF and undergo apheresis either through placement of catheters in antecubital veins or a temporary central venous catheter,
  2. Healthy,
  3. Willing,
  4. For recipients of an unrelated donor transplant, recipient eligibility will be restricted as follows if in the judgment of the recipients' transplant physician, the recipient cannot receive a transplant with combined positive and negative fractions as described in Section 6.1.3.2 or an unmanipulated PBSC product.
  5. Meets eligibility criteria for donors.
* If only one mismatched related relative is available, an acceptable unrelated donor must be identified as a backup.
* Patient or authorized guardian must sign informed consent for this study.

Exclusion Criteria:

* Patient with an anticipated life expectancy of < 1 month
* Active infectious hepatitis or CMV infection
* HIV or HTLV-I/II infection
* Serious infection (bacterial, fungal, viral) within the last 4 weeks
* Cardiac ejection fraction < 45%; can be lower if patient is not in clinical cardiac failure and a reduced intensity conditioning regimen is used.
* Creatinine clearance <60 ml/min/1.72 m2; can be lower if a reduced intensity conditioning regimen is used.
* Pulmonary diffusion capacity (adjusted for Hgb), FEV1, or FVC <60% of predicted or O2 sat < 94% if unable to perform PFTs; can be lower if a reduced intensity conditioning regimen is used.
* Serum ALT > 3 x upper limit of normal (can be up to 5 x upper limit of normal if a reduced intensity conditioning regimen is used) or bilirubin > 2. The bilirubin criteria for sickle cell disease patients is direct bilirubin >2x upper limit of normal.
* Performance score (Lansky/Karnofsky) < 50
* Any condition that compromises compliance with the procedures of this protocol, as judged by the principal investigator.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2009-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Gilman, MD, Principal Investigator — Department of Pediatrics, Levine Children's Hospital, Carolinas Healthcare System
Locations (1):
- Levine Children's Hospital, Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gilman AL, Eckrich MJ, Epstein S, Barnhart C, Cannon M, Fukes T, Hyland M, Shah K, Grochowski D, Champion E, Ivanova A. Alternative donor hematopoietic stem cell transplantation for sickle cell disease. Blood Adv. 2017 Jun 28;1(16):1215-1223. doi: 10.1182/bloodadvances.2017005462. eCollection 2017 Jul 11. PMID 29296761

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Candidates for bone marrow transplant who did not have a healthy HLA-identical related donor, at Levine Children's Hospital between December 2009 and June 2016.
Pre-assignment Details: Subjects were enrolled to two cohorts based on donor type, Mismatched Related Donor (MMRD) and Matched Unrelated Donor (MUD).
Groups:
- T Cell Depletion Using CliniMACS®: Recipients will receive T cell-depleted PBSC from eligible donors after receiving conditioning therapy using CliniMACS® device.
  CliniMACS® (T cell depletion): Stem cells will be collected from donors after they receive Granulocyte colony-stimulating factor (G-CSF). The cells will be processed using the CliniMACS device to select for CD34+ stem cells and to deplete T cells. Recipients will receive conditioning therapy that is based on their disease type and then receive the CD34+ stem cells.
Period: Overall Study
Arm/Group | T Cell Depletion Using CliniMACS®
Started | 53 (One patient, FDA and IRB approved to enroll as an exception, was not evaluable for study endpoints.)
Completed | 52
Not Completed | 1
Not completed — Protocol exception/ not evaluable | 1

BASELINE CHARACTERISTICS:
Arm/Group | T Cell Depletion Using CliniMACS®
Number analyzed (Participants) | 52
Age, Customized [Count of Participants; unit: Participants]
  Less than 1 year | 4
  1-2 years | 3
  2-4 years | 5
  4-6 years | 6
  6-8 years | 3
  8-10 years | 4
  10-12 years | 6
  12-14 years | 5
  14-16 years | 5
  16-18 years | 8
  Greater than 18 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 10
  African American | 26
  Hispanic or Latino | 13
  Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Severe Graft vs. Host Disease (GVHD).
Description: Severe GVHD defined as grade III/IV GVHD.
Time Frame: Within 30 days after stem cell transplant
Measure: Count of Participants; unit: Participants
Arm/Group | T Cell Depletion Using CliniMACS®
Number analyzed (Participants) | 52
Participants | 0

2. Secondary Outcome: Number of Participants With Engraftment and Time to Engraftment
Description: Engraftment was measured as time to absolute neutrophil count >500
Time Frame: Within 28 days after stem cell transplant
Population: There were 2 cases of primary graft failure in the mismatched related donor cohort; both achieved engraftment following a second transplant.
Measure: Mean (Full Range); unit: days
Arm/Group | Mismatched Related Donor Cohort | Matched Unrelated Donor Cohort
Number analyzed (Participants) | 41 | 9
days | 15 [9 to 19] | 13 [10 to 15]

3. Secondary Outcome: Number of Participants With Post-transplant Infections
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | T Cell Depletion Using CliniMACS®
Number analyzed (Participants) | 52
Participants
  HHV-6 reactivation, no disease | 39
  Viral URI (adeno, paraflu, rhino, rsv) | 25
  Clostridium difficile colitis | 24
  Adenovirus reactivation, no disease | 15
  Bacteremia, gram positive | 12
  Candidiasis (not invasive) | 11
  Sinusitis | 11
  Bacteremia, gram negative | 9
  CMV reactivation, no disease | 9
  BK virus, no disease | 7
  EBV-related lymphoproliferative disease | 6
  BK virus, hemorrhagic cystitis | 5
  Adenovirus disease | 5
  Infection with normal ANC - grade 3 | 5
  Norovirus | 5
  Positive Galactomannan | 5
  Acute otitis media | 4
  HSV - mouth sores | 4
  EBV reactivation, no disease | 4
  Pneumonia | 3
  Varicella zoster | 3
  Candidiasis (invasive) | 2
  CMV, GI disease/ encephalitis | 2
  Disseminated aspergillus | 2
  Methicillin-Resistant Staph Aureus | 2
  Rotavirus | 2
  Nocardia | 2
  Pneumonia - fungal (non-aspergillus) | 1
  Influenza | 1
  Parvovirus B19 (low level) | 1
  Sapovirus | 1
  Septic arthritis (prosthetic joint) | 1
  Possible respiratory infection (rhizomucor) | 1

4. Secondary Outcome: Number of Participants With EBV-related Post Transplant Lymphoproliferative Disorder (PTLD)
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | T Cell Depletion Using CliniMACS®
Number analyzed (Participants) | 52
Participants | 6

5. Secondary Outcome: Number of Participants With Post-transplant Leukemia Relapse
Time Frame: 5 years
Population: Of the 43 recipients in the mismatched related donor cohort, 24 of those had leukemia. No recipients in the matched unrelated donor cohort had leukemia.
Measure: Count of Participants; unit: Participants
Arm/Group | T Cell Depletion Using CliniMACS®
Number analyzed (Participants) | 24
Participants | 5

6. Secondary Outcome: Number of Participants With Transplant-related Mortality
Description: Transplant-related mortality includes death due to regimen-related toxicity or GVHD (all causes other than disease relapse). Those who died due to disease relapse are not included in the analyzed population for that time point.
Time Frame: 2 year
Population: Those who died due to disease relapse are not included in the analyzed population for that time point.
Measure: Count of Participants; unit: Participants
Arm/Group | T Cell Depletion Using CliniMACS®
Number analyzed (Participants) | 52
Participants
  Day 100: number analyzed (Participants) | 51
  Day 100 | 1
  1 year: number analyzed (Participants) | 48
  1 year | 9
  2 years: number analyzed (Participants) | 47
  2 years | 11

7. Secondary Outcome: Number of Participants With Transplant-related Toxicities
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | T Cell Depletion Using CliniMACS®
Number analyzed (Participants) | 52
Participants
  Thrombotic Microangiopathy | 8
  Idiopathic Pneumonia Syndrome | 3
  Veno-occlusive Disease | 1

8. Secondary Outcome: Overall Survival
Time Frame: 2 years
Population: Subjects at least 2 years after transplant are evaluable for 2 year overall survival.
Measure: Count of Participants; unit: Participants
Groups:
- Mismatched Related Donor Cohort: Malignant Disease: Number of recipients alive following bone marrow transplant for malignant disease.
- Mismatched Related Donor: Non-malignant Disease; Matched Unrelated Donor Cohort: Number of recipients alive following bone marrow transplant for non-malignant disease.
Arm/Group | Mismatched Related Donor Cohort: Malignant Disease | Mismatched Related Donor: Non-malignant Disease | Matched Unrelated Donor Cohort
Number analyzed (Participants) | 17 | 13 | 7
Participants | 9 | 9 | 6

9. Secondary Outcome: Device Performance: Dose of CD34+ Cells and CD3+ Cells Given
Description: For mismatched related donors, the target cell dose after processing is >/= 20 x 10^6 CD34+ cells/kg patient body weight, but >/= 8 x 10^6 is acceptable.
  For unrelated donors the target cell dose after processing is >/= 10 x 10^6 CD34+ cells/kg patient body weight, but >/= 4 x 10^6 is acceptable.
  The target T cell dose is </= 3 x 10^4 CD3+ cells/ kg.
Time Frame: Length of the trial (5 years)
Measure: Mean (Full Range); unit: cells/ kg
Arm/Group | Mismatched Related Donor Cohort | Matched Unrelated Donor Cohort
Number analyzed (Participants) | 43 | 9
cells/ kg
  x 10^6 CD34+ cells/ kg | 20.26 [8.78 to 25.03] | 15.16 [11.06 to 23.33]
  x 10^4 CD3+ cells/ kg | 0.02 [0 to 1.1] | 0.3 [0 to 0.5]

ADVERSE EVENTS:
Time Frame: From the start of the conditioning regimen for transplant until 1 year after transplant
Arm/Group | T Cell Depletion Using CliniMACS®
All-Cause Mortality (participants affected / at risk) | 15/52
Serious Adverse Events (participants affected / at risk) | 45/52
Other Adverse Events (participants affected / at risk) | 33/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | T Cell Depletion Using CliniMACS® (N=52)
Fever (General disorders) | 32
HHV-6 Reactivation (Infections and infestations) | 9
Graft vs. Host disease (Immune system disorders) | 9
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 6
Acute gastroenteritis/ diarrhea (Gastrointestinal disorders) | 5
CMV reactivation (Infections and infestations) | 4
EBV-related lymphoproliferative disease (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 4
Infection w/ unknown absolute neutrophil count (ANC) (Infections and infestations) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Hemorrhagic cystitis (Renal and urinary disorders) | 3
Relapse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/26
Decreasing donor chimerism (Blood and lymphatic system disorders) | 2
Infection - grade 4 (Infections and infestations) | 2
Seizures (Nervous system disorders) | 2
Viral upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Renal & Urinary disorder - grade 3 (Renal and urinary disorders) | 1
Pneumoatosis Intestinalis (Gastrointestinal disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Mucositis/ dehydration (Gastrointestinal disorders) | 1
Leukopenia/ Neutropenia - grade 3 (Blood and lymphatic system disorders) | 1
Infusion reaction (General disorders) | 1
Hypothermia (General disorders) | 1
Hypertension (Vascular disorders) | 1
Pulmonary/ Upper Respiratory- other (Respiratory, thoracic and mediastinal disorders) | 1 — Blood tinged sputum, following fungal pneumonia
Graft failure (Blood and lymphatic system disorders) | 1
Infection - eye (Infections and infestations) | 1
Dehydration with hypernatremia (Metabolism and nutrition disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T Cell Depletion Using CliniMACS® (N=52)
Hypoxia - grade 3 (Respiratory, thoracic and mediastinal disorders) | 14
Rash - grade 3 (Skin and subcutaneous tissue disorders) | 5
Seizures - grade 3 (Nervous system disorders) | 5
Hypokalemia - grade 4 (Metabolism and nutrition disorders) | 4
Hypoxia - grade 4 (Respiratory, thoracic and mediastinal disorders) | 4
Renal and Urinary disorder - grade 3 (Renal and urinary disorders) | 4
Thrombotic microangiopathy - grade 4 (Blood and lymphatic system disorders) | 4
Thrombotic microangiopathy - grade 3 (Blood and lymphatic system disorders) | 4
Elevated ALT - grade 4 (Investigations) | 3
Hypertension - grade 4 (Vascular disorders) | 3
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 3
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 3
Renal disorder - grade 4 (Renal and urinary disorders) | 3
Thrombosis - grade 3 (catheter-related) (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2015-01-30): https://cdn.clinicaltrials.gov/large-docs/64/NCT00968864/Prot_SAP_000.pdf
  • Informed Consent Form: Recipient Consent (2015-01-30): https://cdn.clinicaltrials.gov/large-docs/64/NCT00968864/ICF_001.pdf
  • Informed Consent Form: Donor Consent (2014-03-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT00968864/ICF_002.pdf